CLINICAL TRIAL: NCT05594433
Title: Donation of Whole Blood by Healthy Volunteers After Mobilisation by Haematopoietic Growth Factor for Validation of a Cell Expansion Automaton Allowing the Simultaneous Production of Several Cell Grafts for Therapeutic Use
Brief Title: Donation of Whole Blood by Healthy Volunteers After Mobilisation by Haematopoietic Growth Factor (Rhu-G-CSF = Granocyte)
Acronym: CARDIOSTEM
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CellProthera (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2013-A01558-37
Record Dates: First submitted 2022-10-13; First posted 2022-10-26 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Lenograstim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Sub cutaneous injection of Lenograstim with blood donation (450ML) after 4 days of mobilization
  Interventions: Drug: Lenograstim

INTERVENTIONS:
Drug: Lenograstim — Injection sub cutaneous of Lenograstim during 4 days, once per day
  Other Names: Granocyte(R)

SUMMARY:
Donation of whole blood by healthy volunteers after mobilisation by haematopoietic growth factor (rhu-G-CSF = Granocyte) for biological validation of a cell expansion automaton allowing the simultaneous production of several cell grafts for therapeutic use in the cardiac field - 2nd STAGE

DETAILED DESCRIPTION:
The rationale for the MHS002 study is based on the expansion results obtained with the first version of the machine (MHS001):

* Average expansion rate of about 20-fold of CD34+ stem cells observed in a reproducible way on the Mulhouse and Créteil sites,
* No significant difference in phenotypic, immunological or morphological characteristics between the "naive" cells (not multiplied) and the cells after multiplication, nor any chromosomal alteration or hyperploidy: the expansion process developed does not lead to any cellular modification,
* Variability in the number of stem cells obtained after multiplication between healthy volunteers.

Developing a second generation prototype capable of producing 15 grafts per month, it is necessary to proceed with its biological validation, in the same way as the first generation prototype (protocol MHS001) was validated, following the requirements of regulatory agencies. Furthermore, in view of these results, it appeared necessary to define the lower limit of the number of CD34+ stem cells composing the graft, below which the therapeutic efficacy will be reduced or nil. This second stage of the study will make it possible to validate a potency test, i.e. a test making it possible to define the composition and potential effectiveness of the graft before its reinjection.

Given the absence of serious adverse events following the administration of G-CSF in healthy volunteers and in the context of the continued development of the second version of the automaton, validations similar to the first protocol are still necessary. Blood donation from healthy volunteers following stem cell mobilisation by G-CSF administration will allow validation of the second version.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers,
* Age ≥ 18 years and ≤ 60 years,
* Agreeing to the collection of blood products by whole blood donation for scientific research purposes,
* Fit for collection by the collecting physician after a medical examination including measurement of blood pressure, heart rate, electrocardiogram and assessment of venous potential,
* Minimum weight: 50 kg,
* Body mass index (BMI) < 30,
* Haemoglobin level between 13 g/dL and 18 g/dL,
* Platelet count between 150.106/mL and 400.106/mL
* White blood cell count ≥ 3.9.106/mL with neutrophils ≥ 2.5.106/mL,
* Agreement to be registered in the national research file,

Exclusion Criteria:

* Any cardiopulmonary abnormality on initial clinical and ECG assessment
* Clinical measurement of systolic BP ≤ 110 mmHg and/or diastolic BP < 70 mmHg on initial workup
* Any blood work-up abnormality deemed significant by the investigator at the time of the initial work-up,
* Previous administration of any haematopoietic growth factor,
* Regular use of medication(s) within 8 days prior to the start of the Granocyte mobilisation phase,
* Any significant cardiovascular history within the last 2 years
* Any history of severe pulmonary disease (including bacterial or viral pneumonia)
* Any history of cancer (solid tumours or haematological malignancies)
* Anysevere neurological history
* Any severe psychiatric history
* Renal history (creatinine clearance from stage 1 to stage 5 of the HAS 2012 classification)
* Twins with a living twin brother or sister,
* Allergy to any of the excipients of Granocyte,
* History of severe drug allergy, anaphylactic allergic shock or angioedema
* Pre-existing splenomegaly
* Obesity (BMI 30),
* Autoimmune diseases,
* Alcohol and drug abuse, drug abuse
* Blood donation within 2 months prior to inclusion
* Volunteer registered or wishing to register on the bone marrow donor list,
* Sickle cell disease,
* Presence of positive virological markers (anti HIV1 and 2, HTLV1 and 2, anti-HCV, anti-HBS, anti-HBC serologies), active syphilis,
* Rheumatoid arthritis,
* Anticoagulant therapy,
* History of cutaneous vasculitis
* Phenylketonuria,
* Subject on exclusion from another study
* Subject under administrative or judicial supervision
* Subject who would receive more than 4500 euros in compensation due to participation in other research in the 12 months preceding this study,

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-09-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of blood donation of CD34+ stem cells obtained to validate the new automaton | From day 0 of mobilization phase to day 5 corresponding to day of blood harvest
  Validation of the second generation of the automaton able to expend CD34+ stem cells, by collection of 450 mL of blood containing CD34+ stem cells. Blood will be collected after 4 days of mobilization with haematopoietic growth factor (rhu-G-CSF = Granocyte)

SECONDARY OUTCOMES:
Number of CD34+ cells obtained with the second generation machine | From Day 0 to Day 9 expansion
  Confirm that the number of CD34+ cells obtained with the "2nd generation" machine is equivalent to that obtained with the 1st generation machine

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Mutter, MD, Principal Investigator — CHRU Strasbourg
Locations (2):
- France (2):
  - GHU La Pitié-Salpêtrière, Paris
  - CHRU Strasbourg, Strasbourg